CLINICAL TRIAL: NCT05971108
Title: Real-world Elecsys® GAAD Algorithm Implementation and Validation to Improve Surveillance and Early Detection of Hepatocellular Carcinoma
Brief Title: Real-world Elecsys® GAAD Implementation and Validation to Improve Surveillance and Early Detection of HCC
Acronym: REVISE-HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other); Roche Pharma AG (Industry); Unity Insights (Unknown); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B01938
Record Dates: First submitted 2023-05-24; First posted 2023-08-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Liver Cirrhosis; Hepatocellular Carcinoma
Keywords: GAAD; hepatocellular carcinoma; cirrhosis; health inequalities; surveillance
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with liver cirrhosis eligible for HCC Surveillance (Experimental): Real-world HCC surveillance cohort will be exposed to Elecsys® GAAD in parallel with standard of care tests.
  Interventions: Diagnostic Test: Elecsys® GAAD

INTERVENTIONS:
Diagnostic Test: Elecsys® GAAD — Elecsys® GAAD is a CE marked in vitro diagnostic (IVD) multivariate index assay, intended as an aid in the diagnosis of early-stage HCC. It provides a semi quantitative result by combining in an algorithm the quantitative measurements of Elecsys® AFP (alpha-fetoprotein) and Elecsys® PIVKA-II (protein induced by vitamin K absence II) levels in serum and plasma, with gender and age. Clinical evidence showed that Elecsys® GAAD had high performance in detecting HCC (sensitivity 86.5%), particularly early stage (sensitivity 78.9%), with 91.4% specificity for both early and all stages, out-performing current standard of care (Chan et al. 2021). Elecsys® GAAD may be integrated into current surveillance practice to increase early-stage HCC detection rate, reduce unnecessary onward investigations and patient anxiety.

SUMMARY:
Patients with liver cirrhosis are at high risk of developing hepatocellular carcinoma (HCC) which implies significant mortality. At present current surveillance methods detect hepatocellular carcinomas at a late stage resulting in few treatment options for patients and, in the majority of cases, premature death.

The goal of this study is to implement Elecsys® GAAD in real-world hepatocellular carcinoma surveillance for those with liver cirrhosis.

The main questions it aims to answer are:

* Does the introduction of the Elecsys® GAAD algorithm to the surveillance pathway increase early detection of HCC?
* Does the introduction of the Elecsys® GAAD algorithm to the surveillance pathway reduce false positive tests and unnecessary confirmatory investigations?
* Does the new surveillance pathway improve adherence?

Researchers will compare Elecsys® GAAD with standard of care tests to see if it results in earlier detection of hepatocellular carcinoma and will explore potential improvements to the surveillance pathway.

ELIGIBILITY:
Inclusion Criteria:

• Patients with known liver cirrhosis referred into or already under hepatocellular carcinoma surveillance

Exclusion Criteria:

* Pregnancy/breast-feeding.
* Patients who do not have liver cirrhosis
* Patients who already have hepatocellular carcinoma
* Any patient who is unable to understand, retain and weigh information to make an informed decision, will be excluded from the study. The investigators will use every opportunity, including tele-interpretation services to minimise this from happening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological sex used in diagnostic algorithm
Enrollment: 600 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hepatocellular carcinoma diagnosis | 2 years
  Incidence recorded as number of cases per study cohort
Stage of hepatocellular carcinoma at diagnosis | 2 years
  Barcelona Clinic Liver Cancer (BCLC) stage 0-D

SECONDARY OUTCOMES:
Rates of false positives for each combination of diagnostic tests | 2 years
  Count (%) of True/False positives for each test (against magnetic resonance imaging (MRI) / computerised tomography (CT)) will be reported.
  Results from different tests (and their (meaningful) combination) will be tabulated against each other:
  * Alpha-fetoprotein (AFP) vs GAAD
  * Ultrasound scan (USS) vs GAAD
  * AFP+ USS vs GAAD
  * AFP+USS vs GAAD +USS
  * AFP/GAAD/USS/AFP+USS/GAAD+USS vs MRI/CT for those who proceed to confirmatory imaging.
Rates of curative treatment | 2 years
  Rates of curative treatment being offered (%) will be recorded on an intention to treat (ITT) basis from Multi-Disciplinary Team (MDT) meeting outcomes.
Rates of adherence | 2 years
  • Attendance rates for biannual surveillance appointments (%), within predefined tolerance of 5-9 months post previous appointment.
Rates of discontinuation | 2 years
  • Count (%) of surveillance discontinuation, defined as no visit >12 months.
Survival rates | 7 years
  Long-term follow up data will be collected to determine rates of survival following HCC diagnosis at 1-year, 3-years and 5-years.

CONTACTS AND LOCATIONS:
Overall Officials: Varinder Athwal, MRCP PhD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No